CLINICAL TRIAL: NCT03440450
Title: A Phase 1 Dose-escalation Study of FF-10832 for the Treatment of Advanced Solid Tumors
Brief Title: A Phase 1 Dose-escalation Study of FF-10832 for Treatment of Solid Tumors Including Biliary Tract Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fujifilm Pharmaceuticals U.S.A., Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FF10832US101
Record Dates: First submitted 2018-02-09; First posted 2018-02-22 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumors; Biliary Tract Cancer
Keywords: Liposomal gemcitabine
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Intervention Model Description: Open label, dose escalation
Masking Description: None, open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1: Treatment at 1.2 mg/m2 (Experimental): FF-10832 Gemcitabine Liposome Injection, 1.2 mg/m2 administered intravenously (IV) on Days 1 and 15 of each 28-day cycle
  Interventions: Drug: FF-10832 Gemcitabine Liposome Injection
- Cohort 2: Treatment at 2.4 mg/m2 (Experimental): FF-10832 Gemcitabine Liposome Injection, 2.4 mg/m2 administered intravenously (IV) on Days 1 and 15 of each 28-day cycle
  Interventions: Drug: FF-10832 Gemcitabine Liposome Injection
- Cohort 3: Treatment at 4.8 mg/m2 (Experimental): FF-10832 Gemcitabine Liposome Injection, 4.8 mg/m2 administered intravenously (IV) on Days 1 and 15 of each 28-day cycle
  Interventions: Drug: FF-10832 Gemcitabine Liposome Injection
- Cohort 4: Treatment at 8 mg/m2 (Experimental): FF-10832 Gemcitabine Liposome Injection, 8 mg/m2 administered intravenously (IV) on Days 1 and 15 of each 28-day cycle
  Interventions: Drug: FF-10832 Gemcitabine Liposome Injection
- Expansion Cohort: Treatment at Recommended Phase 2 Dose (RP2D) (Experimental): For patients with biliary tract cancer: FF-10832 Gemcitabine Liposome Injection, RP2D administered intravenously (IV) on Day 1 of each 21-day cycle
  Interventions: Drug: FF-10832 Gemcitabine Liposome Injection

INTERVENTIONS:
Drug: FF-10832 Gemcitabine Liposome Injection — FF-10832 to be diluted in dextrose 5% in water (D5W) and intravenously infused at a continuous rate over 30 to 120 minutes
  Other Names: FF-10832

SUMMARY:
To determine the safety profile, maximum tolerated dose (MTD), dose-limiting toxicities (DLT) and recommended Phase 2 dose (RP2D) in patients who receive FF-10832 (Gemcitabine Liposome Injection) for treatment of advanced solid tumors including biliary tract cancer

DETAILED DESCRIPTION:
Dose-escalation Phase:

Eligible patients will receive FF-10832 in 28 day or 21 day cycles. Dosing will continue until progression of disease, observation of unacceptable adverse events, intercurrent illness, or changes in the patient's condition that prevents further study participation after discussion between the Investigator and the Medical Monitor. A number of cohorts will be enrolled sufficient to determine the MTD and to identify the RP2D.

Expansion Phase:

One cohort of biliary tract cancer will enroll up to 18 patients in a 21 day cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years of age
2. Histologically or cytologically confirmed metastatic solid tumor, relapsed or refractory to standard therapy, or for which no standard therapy is available that is expected to improve survival by at least three months
3. At least 3 weeks beyond the last chemotherapy (or 3 half-lives, whichever is shorter), radiotherapy, major surgery, or experimental treatment, and recovered from all acute toxicities (≤ Grade 1), prior to the first dose of FF-10832
4. Cohort expansion phase: (biliary tract cancer):

   * Histologically or cytologically confirmed cholangiocarcinoma or gall bladder carcinoma that is metastatic pancreatic adenocarcinoma following progression or relapseor unresectable
   * Measurable disease by RECIST 1.1
   * Progressed on at least one prior regimengemcitabine-cisplatin therapy or gemcitabine-based therapy if unable to tolerate cisplatin. Adjuvant therapy counts as such therapy.
   * Progressed on, declined on, or was ineligible for therapies directed against fibroblast growth factor (FGFR) and/or isocitrate dehydrogenase (IDH) mutations for tumors appropriately treated with such therapies
   * No more than 3 prior systemic therapies for their tumor. Please contact the medical monitor if there are any questions about eligibility.
   * A serum albumin level ≥ 3 g/dL on entry to the study
5. Adequate performance status: Eastern Cooperative Oncology Group (ECOG) ≤ 1
6. Life expectancy of ≥ 3 months
7. Ability to provide written informed consent

Exclusion Criteria:

1. Patients who have not received standard/approved therapies expected to improve survival by at least 3 months
2. Prior hypersensitivity to gemcitabine
3. Known positive for human immunodeficiency virus (HIV), hepatitis B virus surface antigen (HBsAg) or hepatitis C virus (HCV)

7. Active infection requiring intravenous (IV) antibiotic usage within the last week prior to study treatment

8. Any other medical intervention or other condition which, in the opinion of the Principal Investigator, could compromise adherence to study requirements or confound the interpretation of study results

9. Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Determine incidence of Treatment Emergent Adverse Events (TEAE) | 2.5 years
  Safety and tolerability assessed by adverse events (AEs) and serious adverse events (SAEs)
Identify dose-limiting toxicities (DLT) of FF-10832 | 2.5 years
  DLT is defined as any adverse event at least possibly related to FF-10832, and meeting specified DLT criteria
Determine maximun tolerated dose (MTD) of FF-10832 | 2.5 years
  MTD is defined as the next lower dose of a cohort where patients experienced a DLT

SECONDARY OUTCOMES:
Disease Assessment by CT or MRI scan for solid tumors | 2.5 years
  Disease assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST v. 1.1), clinical benefit is defined as best response of complete response (CR), partial response (PR), stable disease (SD) or disease progression (DP)
Disease Assessment by CT or MRI + PET scan for pancreatic cancer | 2.5 years
  For solid tumors assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST v. 1.1), clinical benefit is defined as best response of complete response (CR), partial response (PR), stable disease (SD) or disease progression (DP). European Organisation for Research and Treatment of Cancer (EORTC) criteria will be utilized for PET response assessments.
Duration of Response | 2.5 years
  Duration of Response is calculated from the date of first response to the date of progression or death
Duration of Stable Disease | 2.5 years
  Duration of Stable Disease is the length of time from the start of the treatment until the criteria for progression are met
Time to progression (TTP) | 2.5 years
  Time to progression is calculated from the date of first treatment to the date of first progression
Progression-free survival (PFS) | 2.5 years
  Progression-free survival will be calculated from the date of first treatment to the date of progression or death
Overall survival (OS) | 2.5 years
  Overall survival will be calculated from the date of first treatment to the date of death from any cause; patients who do not experience death will be censored at the last follow-up time.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Honor Health Research Institute, Scottsdale, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - Hoag Memorial Hospital Comprehensive Cancer Center, Newport Beach, California
  - Sarah Cannon Research Institute, Denver, Colorado
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Research Center, Houston, Texas
  - Virginia Mason Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No